CLINICAL TRIAL: NCT04098666
Title: Metformin in Alzheimer's Dementia Prevention
Acronym: MAP
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Aging (NIA) (NIH); University of Rochester (Other); University of Iowa (Other); Boston University (Other); Wake Forest University (Other); Rush University (Other); Pennington Biomedical Research Center (Other); University of Miami (Other); Emory University (Other); Georgetown University (Other); NYU Langone Health (Other); University of California, Berkeley (Other); The University of Texas Health Science Center at San Antonio (Other); University of Washington (Other); State University of New York - Upstate Medical University (Other); University of Texas Southwestern Medical Center (Other); University at Buffalo (Other); University of Cincinnati (Other); Eastern Virginia Medical School (Other); Medical College of Wisconsin (Other); University of Kansas Medical Center (Other); University of New Mexico (Other); Stanford University (Other); University of California, Irvine (Other); Cornell University (Other)
Responsible Party: Principal Investigator, José A. Luchsinger, Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAS6912; R01AG062624 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: randomized 1:1 placebo controlled double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the study will be placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- metformin users (Experimental): Extended release metformin 500 mg tablets up to 2,000 mg (4 tablets) a day once at night. The maximum dose will be attempted during a titration period in the first month of the study.
  Interventions: Drug: extended release metformin
- metformin non-users (Placebo Comparator): Placebo tablets identical to extended release metformin 500 mg tablets up to 4 tablets a day once at night. The maximum dose will be attempted during a titration period in the first month of the study.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Placebo oral tablet — Placebo tablet identical to metformin, up to 4 tablets a day
  Other Names: Placebo
  Arms: metformin non-users
Drug: extended release metformin — Metformin extended release 500 mg tablets, up to 4 tablets a day
  Other Names: Metformin
  Arms: metformin users

SUMMARY:
MAP will be a multisite phase II/III 1:1 randomized controlled trial (RCT) of long acting metformin (reduced mass Glucophage XR) vs. matching placebo in 326 men and women with early and late aMCI, without diabetes, not treated with metformin, overweight or obese, aged 55 years to 90 years. The RCT will last 18 months and have 4 visits: baseline, 6-months, 12-months, and 18-months. The RCT will be preceded by a screening phase followed by randomization and a titration period in which drug/placebo will be titrated from 500 mg a day (one tablet) to 2,000 mg a day (4 tablets), in increments of 500 mg (one tablet) every 10 days. Participants will remain in the RCT on the tolerated dose, and included in analyses on an intent to treat basis. We expect the attrition rate to be 10%/year. Neuropsychological battery, clinical interviews, physical exam, and phlebotomy will be conducted at baseline and every 6 months. Brain MRI will be conducted in approximately half of the participants (186) twice, at baseline, and after the last study visit at month 18. We will also conduct brain amyloid Positron Emission Tomography (PET) using 18F-Florbetaben, and tau PET using 18F-MK6240 in half of the participants at baseline and end of the RCT.

The primary clinical outcome of the study will be changes in the Free and Cued Selective Reminding Test. The secondary endpoints are 1) changes in global cognitive performance, measured with the Alzheimer's Disease Cooperative Study Preclinical Alzheimer Cognitive Composite (ADCS-PACC); 2) changes in neurodegeneration, ascertained as cortical thickness in areas affected by AD on brain MRI; 3) changes in cerebrovascular disease, ascertained as white matter hyperintensities (WMH) volume on brain MRI; 4) Changes in whole brain amyloid ß (Aß) SUVR and in incident amyloid positivity; 5) Changes in tau SUVR in a composite brain region comprising medial and inferolateral temporal cortex; 6) Changes in plasma AD biomarkers.

The data coordinating center and Imaging Core is located at John Hopkins University. The PET coordinating center is located at UC-Berkeley. The Clinical Coordinating and Monitoring Center and the central laboratory will be located at Columbia. The Research pharmacy function will be shared by the University of Rochester, which will dispense randomization kits, and the University of Iowa, which will receive bulk metformin and identical matching placebo from EMD Serono.

DETAILED DESCRIPTION:
STUDY PROCEDURES AT THE LEVEL OF THE PARTICIPANT.

1. Screening. We propose a 2-tier approach for screening, including telephone pre-screening followed by in-person screening. Telephone screening includes questions about inclusion and exclusion criteria including demographics (age, language), medical history, contraindications to metformin, and medications. In-person screening includes consent, in-person anthropometric measurements (height, weight, waist and hip circumference), vital signs (blood pressure and heart rate), EKG, laboratory tests (TSH, RPR, vitamin B12, complete blood count [CBC], basic metabolic panel [BMP], Hepatic panel, Lipid panel, and Hemoglobin A1c [HbA1c]), and the in person-neuropsychological battery that is used to determine aMCI.
2. Baseline/screening study visit. History includes age, handedness, education, occupation and employment history, past medical history, and all medications utilized, including a judgment as to whether they affect cognition (positively or negatively). Referral source is also documented. Psychiatric history, current and past history of depression, current anxiety, alcohol and other substance use, head injury, hypertension, cardiac disease, thyroid disease, other major medical conditions, and surgery are evaluated at screening. A full medical history will be obtained only at screening. Any report of events, or side effects will prompt a full history and physical exam at any visit. Physical exam will be conducted at screening, with particular emphasis on signs of congestive heart failure, pulmonary, liver, or renal disease for contraindications to metformin, and neurologic examination for the presence of neurologic diseases. Vital signs including blood pressure and heart rate will also be ascertained. Standing height will be measured using a stadiometer calibrated in cm. Body weight is measured using a balance beam scale calibrated in kg. With the participant standing, measurements are taken to the nearest 0.1 kg of weight with a balance scale and height without shoes to nearest 0.5 cm, to calculate BMI (weight in k/height in m2). Waist circumference (WC) is measured at the level of the umbilicus. Hip circumference (HP) is measured at the level of maximal protrusion of the gluteal muscles. Resting Blood Pressure (BP) will be measured using an automated oscillometric device, 3 measurements will be obtained at 1-minute intervals in a seated position after 5 minutes of rest. The average of the 2nd and 3rd measurements will be recorded.

   Neuropsychological battery. Total Recall Score of the Free and Cued Selective Reminding Test (FCSRT). The FCSRT is a 16 item word list with visual and auditory presentation that uses semantic cuing to facilitate encoding and retrieval. The test has a score range of 0 to 48. Paragraph Recall on the Logical Memory IIa (episodic memory): Free recall of 1 short story that consists of 25 bits of information will be elicited immediately after it is read aloud to the subject and again after approximately 30-minute delay. The total bits of information from the story that are recalled immediately (maximum score = 25) and after the delay interval (maximum score = 25) are recorded. The delay score (0-25 story units) will be used in the composite. Digit-Symbol Substitution Test: The Digit Symbol Substitution test is a subset from the WAIS-R. The test consists of 110 small blank squares presented in 7 rows with 1 of 9 numbers (1-9) randomly printed directly above each blank square. A "key" is printed above the rows of blank squares. The "key" pairs numbers 1 through 9 with an unfamiliar symbol. The subject must work as fast as possible for 90 seconds. The measure of interest is number of squares filled in correctly within the time limit (maximum raw score = 110). Mini Mental Status Exam (MMSE). The MMSE scale evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy 2 overlapping pentagons. The MMSE is scored as the number of correctly completed items with a lower score indicative of poorer performance and greater cognitive impairment. The total score ranges from 0 (worse) to 30 (perfect). Trail-Making Test, Part A: This test of visuoperceptual ability, attention and speed consists of 25 circles distributed over a white sheet of 8 1/2" X 11" paper that are numbered. The participant is instructed to connect the circles with a pencil line as quickly as possible all numbers in an ascending order (e.g., 1 to 2; 2 to 3; etc). The participant's performance is judged in terms of the time (in seconds) required to complete the task and by the number of errors of commission and omission. The time to complete the trial will be the measures of interest. Trail-Making Test, Part B: This test of visuoperceptual ability, attention and set-shifting ability consists of 25 circles distributed over a white sheet of 8 1/2" X 11" paper that are either numbered (1 through 13) or contain letters (A through L). The participant is instructed to connect the circles with a pencil line as quickly as possible while alternating between numbers and letters in an ascending order (e.g., A to 1; 1 to B; B to 2; 2 to C). The participant's performance is judged in terms of the time (in seconds) required to complete the task and by the number of errors of commission and omission. The time to complete the trial will be the measures of interest. Trail-Making Test, Part B is available in multiple forms of equal difficulty for purposes of repeated evaluations. ADAScog12. This test will be used as part of the core battery and assesses memory, reasoning, naming, orientation, ideational praxis, constructional praxis, spoken language, language comprehension, word finding difficulty, and ability to remember test instructions. The addition of a 10 word delay recall adds sensitivity in aMCI and yields maximum score of 80. Functional abilities: ADCS-ADL-PI:The ADCS-ADL-PI was developed in the ADCS Prevention Instruments Trial. The subject rates his/her performance of 18 IADL tasks over the past 2 months. Questions about use of technology (e.g., computers and cell phones) are included. Responses for each IADL include improved IADL performance (fewer errors, faster completion, less need to refer to notes or instructions), no change ('as well as usual'), various levels of impaired performance, and non-performance. Clinical Dementia Rating (CDR). The CDR is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively). The score is based on interviews with the subject and study partner, using a structured interview that assesses 6 domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The ratings of degree of impairment obtained on each of the 6 categories of function are synthesized into 1 global rating of dementia (ranging from 0 to 3), with more refined measure of change available by use of the Sum of Boxes (CDR-SB). Reliability and validity has been established, as has high inter-rater reliability. Memory Complaint Questionnaire (MAC-Q): The MAC-Q consists of six items. The first five items relate to specific situations that are frequently reported as troublesome for those with declining memory, and the last item broadly measures overall self-perceived memory decline. Cognitive diagnoses. The research physician will complete the National Alzheimer's Coordinating Centers (NACC) Assessment and Uniform Data Set (UDS), which takes 35 minutes and includes detailed medical and family history, and neurological exam, including the Unified Parkinson's Disease Rating Scale for extrapyramidal signs, psychiatric assessment with the short version of the Geriatric Depression Scale and Neuropsychiatric Inventory (NPI) questions, assessment of vascular risk factors plus the Hachinski scale, and a Clinical Dementia Rating (CDR). Cognitive diagnosis will be examined for inclusion and exclusion purposes and will also be examined as an exploratory outcome. For cognitive diagnosis transitions (i.e. conversion from MCI to dementia), an adjudication panel at the CCMC will conduct monthly consensus meetings or calls. This panel will be comprised of co-investigators Luchsinger, Goldberg, Devanand. During the meeting information of all the cognitive, functional and other clinical information of the subjects will be presented, blind to study allocation. Evidence of cognitive deficits (based on the neuropsychological scores), evidence of impairment in social or occupational function (as assessed by the functional measures), and evidence of cognitive and social-occupational function decline will be the criteria used for the diagnosis of dementia.
3. Randomization. Eligible participants will be randomized in 1:1 ratio to receive either metformin or placebo, using randomly permuted block randomization of size two or four by each site to achieve balance of treatment assignment overall and by site.
4. Titration. After participants consent, are deemed eligible, and complete the baseline assessment, they will complete a 30-day titration period in which the metformin/placebo dose will be increased from 500 mg a day at randomization in increments of 500 mg every 10 days to a maximum of 2,000 mg a day. Participants will have in person visits every 10 days to check on their drug/placebo tolerance.The metformin tablets are taken together as a single dose, usually recommended once at night. Participants will remain on the highest dose tolerated.
5. Baseline Brain MRI. Participants will be invited to have a baseline brain MRI without contrast. We expect that brain 3T MRI will be conducted in 186 participants across all sites. MRI sequences will include 3Plane Gradient Echo Localizer, 3D MPRAGE T1, 3D T2, DTI 30 direction, DTI 30 direction, pCASL Axial, pCASL Axial Calibration. Acquisition of these sequences will take approximately 50 minutes.
6. Baseline Brain Amyloid PET: Amyloid PET imaging will be obtained using 18F-Florbetaben. 18F-Florbetaben will be injected as 8.1 mCi, with image acquisition 90-110 min post injection (following CT or transmission scan) as 4 x 5 min frames.
7. Baseline Tau PET: Tau PET acquisition will entail injection of 10 mCi of MK6240 with imaging from 90-110 min after CT or transmission scan.1086. Monthly and ad-lib follow-up calls, text messages, or mails. We will conduct monthly follow-up calls to inquire about adverse events and issues with metformin tolerance. We will use the ADCS Adverse Event Checklist to monitor adverse events.
8. Follow-up visits: We will repeat all clinical (non-brain imaging) assessments at months 6, 12, and 18. The only exception is that we will test TSH and RPR only at baseline. All other laboratory tests will be repeated. Pill counts will be conducted to assess compliance with metformin and placebo. We will administer the adverse events checklist. All remaining study drug or placebo will be retrieved to assess compliance and for disposal.
9. Follow-up Brain MRI. Participants who undergo a baseline MRI will be invited to have a follow-up brain MRI with the same sequences after the completion of the last visit at month 18. The MRI will be completed within one month of the last visit.
10. Follow-up Brain Amyloid PET: Participants who underwent baseline amyloid PET will be invited to repeat the PET at 18 months.
11. Follow-up Tau PET: Participants who underwent baseline Tau PET will be invited to repeat the PET at 18 months.
12. Monthly and ad-lib follow-up calls, text messages, or mails. We will conduct monthly follow-up calls to inquire about adverse events and issues with metformin tolerance.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of aMCI: in general, the diagnosis of aMCI follows the definition in the 2011 National Institute on Aging (NIA)/ Alzheimer's association (AA) guidelines, without biomarkers. Participants must have:

* Subjective memory concerns reported by participant, study partner, or clinician.
* A mini-mental state exam between ≥ 22 for subjects with more than 8 years of education. For subjects with less than 8 years of education, a MMSE ≥ 20 will be allowed.
* Clinical Dementia Rating = 0.5. The memory box score must be at least 0.5. Information from the formal University of Washington CDR instrument, report by the participant of subjective cognitive complaints, and findings from the screening neuropsychological battery, can be used for this determination by the investigative team. For example, the University of Washington CDR can be 0, but the CDR memory box score can be deemed to be 0.5 based on cognitive complaints at screening and meeting the MCI neuropsychological criteria.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit.
* Abnormal memory function documented by scoring within the education adjusted ranges on the Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised.

  * For early MCI:

    * 9-11 for 16 or more years of education
    * 5-9 for 8-15 years of education
    * 3-6 for 0-7 years of education
  * For late MCI

    * ≤ 8 for 16 or more years of education
    * ≤ 4 for 8-15 years of education
    * ≤ 2 for 0-7 years of education
* Age range: 55 years to 90 years.
* Sex distribution: all eligible men and women will be included and no one will be excluded because of gender.
* Languages: fluent in English or Spanish. We have reliable, well-validated Spanish tests for all outcome measures.
* Participants without a known history of diabetes. If diabetes is diagnosed during screening (hemoglobin A1c of 6.5 % or greater) they will also be excluded. The main justification for this exclusion is the potential for these participants to be placed on other diabetes medications that may confound our study.
* General cognition and functional performance such that a diagnosis of dementia cannot be made at the time of screening based on DSM-V criteria.
* Vision and hearing must be sufficient for compliance with testing procedures.
* Must have an informant to come to all appointments or be available by telephone at follow-up visits.

Study Partner Inclusion Criteria

* The study partner can provide an independent evaluation of functioning for a person enrolled in the MAP study as a participant
* The study partner agrees to attend study visits with the MAP participant or be available by telephone.

Exclusion Criteria:

* Use of metformin or any class of medication approved for treatment of diabetes, even if it is used for an indication other than diabetes (e.g., obesity), within one year of screening. These medications include GLP-1 agonists used for weight loss.
* Body mass index ≤ 20 k/m2.
* Metformin is contraindicated in persons with an estimated glomerular filtration rate (eGFR) of less than 30 mL/min. For persons with an eGFR of 30 to 45 mL/min, a reduction of the dose or discontinuation of the medication is recommended for those on metformin; in this range, it is also recommended that persons do not initiate metformin. Thus, participants with eGFR ≤ 45 mL/min will not be eligible to participate.
* The risk of lactic acidosis is increased in persons with liver disease and class III or IV congestive heart failure. Thus, persons with liver disease other than non-alcoholic fatty liver disease or class III or IV congestive heart failure will not be eligible to participate due to the risks of side effects.
* A history of intolerance to metformin.
* History of cerebrovascular accident with residual neurological deficits.
* Moderate to severe depression, indicated by a score in the Geriatric Depression Scale of 9/15 or higher.
* Dementia diagnosis
* Lack of capacity to consent
* Participants with neurologic diseases associated with neurologic deficits on clinical examination.
* Participants with other current Axis I psychiatric diagnoses such as bipolar disorder or schizophrenia.
* Alcohol or substance abuse or dependence in the past 6 months.
* Use of medications rated as being the likely cause of cognitive impairment. These include benzodiazepines in dose equivalents greater than 2 mg daily of lorazepam, and regular use of prescription narcotics.
* Normal individuals without cognitive complaints.
* Participants with uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg).
* Participants with active cancer or a history of cancer within the last two years, with the exception of squamous or basal cell carcinoma of the skin.
* Participants who for any reason may not complete the study as judged by the study physician.
* Participants planning to move to another city or state during the duration of the study.
* Participants with a known history of diabetes. The rationale for this exclusion is persons with diabetes may already be on metformin or on other medications that increase insulin levels and could confound the trial.
* Participants with diabetes discovered on screening based on American Diabetes Association criteria using HbA1c (HbA1c of 6.5% or greater). Although metformin could be a first treatment of diabetes for these participants, addition of treatments for diabetes by physicians could confound the study.
* Use of any other amyloid modifying treatment for AD such as lecanemab, either experimental or approved by the Food and Drug Administration, is exclusionary. Previous use of amyloid targeting therapy that was shown to be non-efficacious (e.g., solunazemab) is not exclusionary.
* Not able to undergo phlebotomy as reported by the participant or determined by the study coordinator or physician.
* Participants with known, suspected, or plan for becoming pregnant.
* The presence of a medical condition, and/or use of a medication and/or any substance, individually or in aggregate, that in the judgement of the study team, is the primary cause of cognitive impairment. For example, if hypothyroidism, cobalamin deficiency, or tertiary syphilis are reported or found during screening, they could be deemed as being likely contributors to cognitive impairment, and thus be exclusionary. Combinations of multiple medications with anti-cholinergic effects with or without other central nervous system depressants could also be considered as being causative of cognitive impairment and exclusionary.

Exclusion Criteria for MRI

Contraindications for MRI include inability to lie flat, claustrophobia, or presence of indwelling metal objects or implants that are not MRI compatible.

Exclusion Criteria for PET

History of adverse reactions to radiocontrast agents.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Free and Cued Selective Reminding Test (FCSRT) | 18 months
  Total recall of the FCSRT

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study Preclinical Alzheimer's Cognitive Composite (PACC-ADCS) | 18 months
  Composite of 4 tests:The FCSRT, 2. The Delayed Recall score on the Logical Memory IIa subtest from the Wechsler Memory Scale, The Digit Symbol Substitution Test score, from the Wechsler Adult Intelligence Scale-Revised, and the Mini Mental Status total score.
APOE-ε4 genotype | 18 months
  APOE-ε4 genotype as a modifier of the efficacy of metformin
White matter hyper intensity volume (WMH) | 18 months
  total WMH volume adjusted for cranial size
Brain amyloid | 18 months
  Changes in whole brain Amyloid beta standardized uptake value ratio (SUVR) and in incident amyloid positivity. Brain amyloid will be ascertained using 18F-Florbetaben
Brain Tau | 18 months
  Changes in tau SUVR in a composite brain region comprising medial and inferolateral temporal cortex. Tau will be measured using 18F-MK6240
plasma AD biomarkers | 18 months
  Changes in plasma AD biomarkers
Cortical Thickness | 18 months
  Cortical thickness in areas affected by Alzheimer's disease from 3T MRI

CONTACTS AND LOCATIONS:
Overall Officials: José A Luchsinger, MD, Principal Investigator — Columbia University
Locations (22):
- United States (22):
  - University of California - Irvine, Irvine, California
  - Stanford University, Palo Alto, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Wichita, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Boston University, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - University at Buffalo, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cornell University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All datasets used/generated on the project will be made accessible and reusable by qualified individuals other than the original data generators via web-based resources with the capacity to store large and diverse datasets (such as data about clinical phenotypes, genetics, epigenetics, proteomics, and metabolomics) to enable multiple parallel approaches to data analysis and interpretation. All analytical methodologies will be made fully reproducible and transparent so that results can be vetted and existing analysis techniques quickly applied to new application areas. We will comply with the data sharing arrangement decided by NIA.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After reporting of main results

REFERENCES:
- [Derived] Kim AB, Arvanitakis Z. Insulin resistance, cognition, and Alzheimer disease. Obesity (Silver Spring). 2023 Jun;31(6):1486-1498. doi: 10.1002/oby.23761. PMID 37203336

DOCUMENTS (2):
  • Study Protocol (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04098666/Prot_000.pdf
  • Informed Consent Form (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04098666/ICF_002.pdf